CLINICAL TRIAL: NCT04032678
Title: A Comparison of Biphasic Truncated Exponential and Pulsed Waveforms for Cardioversion of Atrial Fibrillation
Brief Title: Comparison of Efficacy and Safety of Two Biphasic Defibrillators in Cardioversion of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University National Heart Hospital (Other)
Responsible Party: Principal Investigator, Elina Trendafilova, Prof., University National Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P4/10.07.2018
Record Dates: First submitted 2019-07-12; First posted 2019-07-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Atrial Fibrillation; Arrythmia; Electric Countershock
Keywords: Cardioversion; Cardiac Arrythmias; Myocardial Injury; Defibrillators; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: This will be a prospective randomized trial (alternating design) where eligible patients will be randomized to treatment with two different defibrillators. Following the order of patient admittance in ICCU-NCH, the attending cardiologist will assign the odd and even eligible patients to the defibrillators in arm 1 and arm 2, respectively. The cardiologist cannot control the order of patient admittance in ICCU-NCH. The alternative randomization design will equalize the number of subjects on each treatment. This study is not designed to control for sex, age, comorbidity, type of device used for cardioversion, cumulative energy delivered during shocks, number of shocks administered. Randomization is performed to limit these and any other confounding factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (DGT7) (Experimental): Cardioversion with a pulsed biphasic waveform Cardioversion is performed by a pulsed biphasic (Multipulse Biowave®) waveform (Schiller Defigard Touch 7 - DGT7, Schiller Medical, France) with recommended by the manufacturer adult pads (FRED-PA1, Schiller) following an energy protocol of 3 consecutive shocks with constant selected energy: 200J, 200J, 200J. The protocol is stopped at successful cardioversion (sinus rhythm at 1 minute post-shock), otherwise after the 3rd shock. Primary endpoint: The cumulative energy delivered by the consecutive defibrillation shocks during cardioversion.
  Other Name: DGT7
  Interventions: Device: Schiller Defigard Touch 7 - DGT7, Schiller Medical, France
- 2 (LP15) (Active Comparator): Cardioversion with a biphasic truncated exponential waveform Cardioversion is performed by a biphasic truncated exponential waveform (LIFEPAK 15, Physio-Control Inc., Redmond, WA, USA) with recommended by the manufacturer adult pads (Redipak QUICK COMBO, Physio-Control) following an energy protocol of 3 consecutive shocks with constant selected energy: 200J, 200J, 200J. The protocol is stopped at successful cardioversion (sinus rhythm at 1 minute post-shock), otherwise after the 3rd shock. Primary endpoint: The cumulative energy delivered by the consecutive defibrillation shocks during cardioversion.
  Other Name: LP15
  Interventions: Device: LIFEPAK 15, Physio-Control Inc., Redmond, WA, USA

INTERVENTIONS:
Device: Schiller Defigard Touch 7 - DGT7, Schiller Medical, France — Cardioversion with a pulsed biphasic waveform
  Arms: 1 (DGT7)
Device: LIFEPAK 15, Physio-Control Inc., Redmond, WA, USA — Cardioversion with a biphasic truncated exponential waveform
  Arms: 2 (LP15)

SUMMARY:
Background: Biphasic truncated exponential (BTE) waveforms are standard for cardiac defibrillation and synchronized cardioversion up to date. BTE waveforms differ by design characteristics and technologies for pulse commutation (rectilinear, standard truncated exponential, pulsed). Clinical evaluation of BTE waveforms can be planned during cardioversion (CVS) as a well-established procedure of atrial fibrillation patients who are able to give consent and also present a more controlled population.

Scarce studies have been found to present the relative efficacy and safety of different BTE waveforms during CVS. The validity of significantly deviating results of the pulsed waveform in one CVS study is questionable.

Objective: To compare the CVS efficacy and safety two different biphasic defibrillators - a standard truncated exponential waveform and a pulsed biphasic waveform.

Experimental design: Patients will be recruited at the Intensive Cardiology Care Unit (ICCU), Cardiology Clinic, University National Heart Hospital (NHH), Sofia, Bulgaria, underwent the pre-CVS medical exams and check for eligibility. All eligible patients will sign a written informed consent prior to the CVS and will receive the standard hospital procedures during CVS, accepted in the NHH, and approved by the NHH Local Ethic Committee.

Atrial fibrillation patients will be alternatively randomized to CVS using one of the two defibrillators, following the same energy selection protocol in both defibrillators. The statistical power analysis will consider a non-inferiority comparison between the cumulative energy actually delivered by both defibrillators.

The secondary CVS outcome measures are: the cumulative success rate (measured at 1 minute post-shock) and number of delivered shocks. Delivered energy will be measured during each shock with a dedicated pulse recording device (approved by the NHH Local Ethic Committee). Heart rhythm will be monitoring in continuously recorded peripheral ECG.

The secondary CVS safety outcome measures: Biochemical markers for myocardial necrosis (high sensitive troponin I - hsTnI, creatine kinase MB fraction - CK-MB) will be evaluated on blood samples taken before and 12 hours after cardioversion; ST-segment changes will be measured in lead II (baseline and 10 s post-shock) and 12-lead ECG; Complications after cardioversion will be measured during 2 hours follow-up period in the ICCU.

DETAILED DESCRIPTION:
Background:

External defibrillators are routinely used for treatment of lethal ventricular arrhythmias (defibrillation) as well as atrial and non-lethal ventricular arrhythmias (synchronized CVS). Commercially available defibrillators generate direct current (DC) shock with various waveforms using distinct technologies. These waveforms are suggested to have different efficacy and safety, aiming at a positive effect with lower cumulative energy, smaller number of shocks, and less post-shock complications and myocardial injury. Therefore, the efficacy and safety of different waveforms has been an object of continuous interest and clinical investigations over the last years. Although the superiority of biphasic over monophasic waveforms is well established, the relative efficacy and safety of the available biphasic waveforms is not clear.

Most defibrillator manufacturers use the biphasic truncated exponential (BTE) waveform. Almost all BTE defibrillators are embedding the impedance compensation technology, which adapts the pulse duration for proper delivery of the selected energy. However, various pulse commutation concepts produce differently shaped waveforms:

* rectilinear (impedance compensation with constant pulse duration);
* standard truncated exponential (impedance compensation with constant tilt);
* pulsed (impedance compensation with constant duty cycle and constant tilt). Clinical studies with patients presenting with shockable life-threatening arrhythmias are difficult to perform for ethical and practical reasons. Several studies have therefore included patients requiring elective CVS for atrial arrhythmias, who are able to give consent and also present a more controlled population. Elective CVS is a standard treatment for patients with atrial arrhythmias and is performed as a day case procedure under general anesthesia. The investigator's bibliographic research found 6 studies from which the dose-response curves of 4 rectilinear, 7 standard truncated exponential and 3 pulsed waveforms have been drawn. Although the major disparities between the studies (success accounted at different delays after CVS, rhythm inhomogeneity, different population sizes, different selected energy levels, etc.) the dose-response curves concentrate within 85-95% success rate and 300-500 joules (J) cumulative energy. More data on the efficacy of the pulsed waveform during CVS are needed.

Various BTE waveforms apply different potential gradients on the thorax that might produce various defibrillation effects. Apart from efficacy, the most important aspect is the patient safety, considering that larger potential gradients in the myocardium lasting longer could potentially induce an electroporation and then a fibrillation. A frequently observed effect of electroporation are the post-shock ST-segment deviations in the surface ECG, representing the potential difference between the normal tissue and sustained depolarized critical mass of myocardium closest to the associated origin of the electrical current. Although ST-segment changes are an easily ignored phenomenon, occurring acutely and resolving during the first few minutes post-shock, their presence in a short-term basis can identify electroporation by dangerously high potential gradients, while the sustained ST-changes in a long-term basis can identify cases with myocardial injury. The most reliable quantification of shock-induced myocardial injuries is based on measurements of the hsTnI biomarker after CVS. The safety of shocks contemplates any other complications after CVS, such as apnea, arrhythmias, etc. The variety of safety outcomes for different BTE waveforms is not clear.

Considering that little published data are available on pulsed waveforms, this study aims to compare the pulsed biphasic waveform to a standard truncated exponential waveform in respect of efficacy and safety in elective CVS of atrial fibrillation.

Methods:

Study population All patients admitted for elective CVS of atrial fibrillation (AFIB) in ICCU- National Heart Hospital (NHH) will be potentially eligible for the study. Informed consent will be obtained from all eligible patients prior to CVS. Patients declining to participate in the study will receive treatment according to the hospital protocol.

Cardiologists in ICCU-NHH will check the eligibility of each patient following the detailed list of inclusion and exclusion criteria in section Eligibility Criteria, based on the documented pre-treatment data (duration of AFIB, concomitant diseases, thyroid dysfunction, transesophageal echocardiographic (TEE) measurements).

Additionally, eligibility will be verified through pre-CVS medical exams and routine blood test within 24 hours before CVS, including hsTnI measurements on the day of CVS:

Study design A prospective randomized trial (alternating design) where eligible patients will be randomized to treatment with two different defibrillators. Following the order of patient admittance in ICCU-NHH, the attending cardiologist will assign the odd and even eligible patients to the defibrillators in arm 1 and arm 2, respectively. The cardiologist cannot control the order of patient admittance in ICCU-NHH. The alternative randomization design will equalize the number of subjects on each treatment. This study is not designed to control for sex, age, comorbidity, type of device used for CVS, cumulative energy delivered during shocks, number of shocks administered. Randomization is performed to limit these and any other confounding factors.

Patient preparation Patients will be consulted prior to CVS in a quiet setting. Any questions will be answered by the attending cardiologist. Patients will be asked to manually sign their informed consent for study participation before further preparations and data collection. If the patient declines to participate, then he/she will receive treatment according to the hospital protocol without data documentation, as further defined in the study.

Demographic data (hospital file ID, age, gender, weight, height, body mass index, body surface area) will be taken.

Pre-treatment data will be read from the patient dossier:

* All concomitant diseases.
* All medications during the previous 7 days before CVS.
* Left atrium dimensions, left ventricle dimensions and volumes, ejection fraction (EF) by transthoracic echocardiography during the last month.
* TEE will be performed for all patients within 1 to 5 days before CVS (except if contraindications of TEE exist); presence of cardiac thrombus and spontaneous echo contrast will be checked.
* Duration of index AFIB in days.
* European Heart Rhythm Association (EHRA) class score of symptoms from index AFIB
* American Society of Anaesthesiologists Score (ASA)
* Signs of heart failure before CVS and on the day before CVS. Standard blood test (taken 24h before CVS) will be documented. Appropriate standard anticoagulation with unfractionated heparin (UFH) or acenocoumarol or direct oral anticoagulants (DOAC) is to be applied before and after CVS.

The patient will be in fasting condition before CVS. If needed, the chest will be shaved before CVS so that the self-adhesive defibrillation pads can be stick intact to the skin.

The anesthesia will be conducted by an anesthesiologist with slow intravenous injection of Propofol, adjusted individually to reach deep sedation. The individual Propofol dose (mg per kg bodyweight) will be documented.

CVS protocol:

The CVS procedure is performed in ICCU by a cardiologist and anesthesiologist. Defibrillator pads are placed according to the manufacturer user guides. Standard self-adhesive defibrillation pads, recommended by specific defibrillator's manufacturer will be used.

Defibrillator use: The time-interval interval between consecutive shocks is ≥ 1 minute; The energy of consecutive shocks follows pre-defined protocol; The protocol stops at successful CVS (sinus rhythm at 1 minute post-shock), otherwise at the last shock of the protocol.

Data collection and Follow up:

* Defibrillator pulse recorder: The shock waveforms delivered by the studied defibrillators is recorded in real-time during the shock by a dedicated measurement recorder (Defimpulse) connected in the patient circuit. This allows accurate measurement of the delivered energy, which is the primary measured outcome. Additionally, currents, voltages, patient impedances at each shock can be also measured. The device is fully automatic and expert assistance is not needed during the CVS intervention. The use of the Defimpulse has been approved by the NHH Ethical Committee.
* Blood samples, standard 12-lead ECG, blood pressure and heart rate is obtained at baseline.
* Continuous ECG in 3 peripheral leads (I, II, III) is recorded during the CVS procedure. ST-segment deviation is measured on the first cardiac complex after 10 s post-shock 80 ms after J point in lead II.
* Standard 12-lead ECG is recorded (5 minutes) after CVS; 24 h after CVS; at discharge if the discharge day is different from 24 h after CVS.
* Heart rate and blood pressure are measured 3 times after CVS (immediately, 1 hour and 2 hours after the last shock).
* Follow-up period in ICCU (2 hours of duration): Potential complications after CVS are recorded:

  1. Presence of apnea
  2. Presence of arrhythmias.
  3. Record of any other medication at CVS and during the follow-up period.
* Follow-up period in the Cardiology Clinic (24 hours of duration):

  1. blood samples to analyze CK-MB and hsTnI (12 hours +/- 4 hours after CVS).
  2. Clinical exam with heart rate and blood pressure: 2 times on the day of CVS.
  3. ECG and blood pressure on the next day after CVS.
  4. Any complications before discharge.

Statistics:

Primary endpoint: The statistical analysis is designed for a non-inferiority comparison between the two defibrillators in respect of their cumulative energies actually delivered. A non-inferiority margin of 50J is chosen as the absolute difference in cumulative delivered energy at the end of the CVS study. It is estimated that a total of 62 patients (31 per group) allows a study power to show non-inferiority of 80%, with a one-sided type I error rate of 0.05.

Continuous variables (cumulative energy, number of shocks, cardiac troponin levels, etc.) will be expressed as mean value ± standard deviation or median values (inter-quartile range) and compared with Students t-test or equivalent non-parametric test, respectively. Categorical variables (e.g. cumulative success rate) are expressed as percentages and compared using the Chi-square or Fisher's exact test (where appropriate). P ≤ 0.05 is considered statistically significant for all comparisons.

Ethics All patients are signed a written informed consent prior to the CVS and receive the standard hospital procedures during CVS, accepted in the NHH and approved by the NHH Ethical Committee. Both defibrillators included in this study are approved for clinical use and both are used on a daily basis.

Data anonymization policy is respected. In order to ensure the medical confidentiality, no information about the patient (intervention place and date, age, gender, name, diagnosis, etc.) is entered in the defibrillators. An identification number are given to each patient by the dedicated measurement recorder (Defimpulse). This number and the recording data are properties of the principal investigator. Approval from the NHH Ethical Committee concerning the use of the Defimpulse during the CVS intervention has been obtained.

ELIGIBILITY:
Inclusion Criteria:

(indications for elective cardioversion of atrial fibrillation):

Patients > 18 years old and:

* Symptomatic AFIB with a duration of less than 12 months - EHRA score 2-4
* Symptomatic first detected AFIB - EHRA score 2-4
* Persistent AFIB after successful causal therapy

Exclusion Criteria:

* The patients are excluded if one of these conditions is present:

  * Patients with atrial flutter
  * Spontaneous HR <60/min
  * Digitalis intoxication
  * Impossibility to maintain sinus rhythm irrespective to antiarrhythmic therapy and frequent cardioversions
  * Conduction disturbances (without fascicular block and AV block 1 degree) in patients without pacemaker
  * Asymptomatic patients with AFIB for > 1 year
  * Thyroid dysfunction: euthyroid status of at least one month is required (TSH is measured).
  * Thrombosis in cardiac cavities, assessment performed using Transesophageal echocardiography (TEE)
  * Spontaneous echo contrast > 2 degree (TEE)
  * Patients with planned cardiac operation in the next three months
  * Patients with embolic event in the last three months
  * Patients <18 years of age
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Defibrillator Efficacy - The cumulative delivered energy | At the end of CVS. Delivered energy (Joules) will be measured during each shock with a dedicated pulse recording device
  The cumulative delivered energy by consecutive defibrillation shocks during cardioversion.
  The cumulative delivered energy is the sum of energies delivered by the consecutive shocks, showing the total energy delivered to the body during cardioversion. It is proportional to the total dissipated heat in the heart that is assumed as the major factor for myocardial injury. The cumulative delivered energies of the two defibrillators will be compared.

SECONDARY OUTCOMES:
Defibrillator Efficacy - The cumulative success rate | At the end of CVS. Peripheral ECG will be continuously recorded during cardioversion and the presence of sinus rhythm will be read by a cardiologist at the first minute after each shock
  The cumulative success rate by the consecutive defibrillation shocks during the cardioversion procedure. The cardioversion success is defined as the conversion of sinus rhythm for at least 1 minute after the shock.The success rate measures the proportion of patients in sinus rhythm one minute after each consecutive defibrillation shock. The cumulative success rate is measured at the final cardioversion shock and defines the final cardioversion outcome. The cumulative success rates of the two defibrillators will be compared.
Defibrillator Efficacy - Number of shocks | At the end of CVS. During the whole cardioversion procedure, each electrical shock delivered to the patient will be counted
  The number of shocks counts the number of delivered consecutive shocks during cardioversion. The maximal number of shocks cannot exceed the number defined in the energy protocol. Less shocks are usually associated with shorter duration of the cardioversion procedure, therefore, preferable in respect of reducing the anesthesia dose, the trauma effect for the patient, and the medical staff employment-time. The number of shocks delivered by both defibrillators will be compared.
Defibrillator Safety - Changes in the concentration of biochemical markers | 12 hours after CVS +/- 4 hours. The blood samples will be taken before cardioversion (on the same day) and after cardioversion (from 8 to 12 hours after the intervention)
  Changes in the concentration of biochemical markers for myocardial necrosis including CK-MB and hsTnI before and after the cardioversion procedure. All blood test are done by hospital clinic of clinical laboratory. Changes in the concentration of hsTnI and CK-MB (post-cardioversion - pre-cardioversion) will be compared between the two defibrillators.
Defibrillator Safety - Complications after cardioversion | 2 hours after CVS. ECG and close patient attendance will be applied during 2 hours follow-up period in Intensive Cardiology Care Unit
  The following post-cardioversion complications will be measured:
  1. Presence of apnea
  2. Presence of arrhythmias, bradycardia or electrical conduction disturbances and the need for their medication during the electrical cardioversion procedure and 2 hours later by continuous ECG monitoring.
Defibrillator Safety - ST-segment changes | At the end of CVS. ST-segment will be measured by a cardiologist in the continuously recorded lead II (immediately before cardioversion and 10s after each shock (80 ms after J point in the first QRS at 10 s post-shock); as well as in standard 12 lead ECG
  ST-segment changes after cardioversion is usually a transient short-lived phenomenon, being maximal just after the shock with a mean duration of 1 minute, and usually resolving 5 minutes post-shock. It is rather associated with electroporation (sustained depolarization of a critical mass of myocardium closest to the associated origin of the electrical current) than with a coronary spasm (leading to transient myocardial ischemia or infarction). The measurement of the ST-shift (mm) and the ST-shift type (depression, elevation) will give a view on the shock-induced electrical potential difference between the depolarized and normal tissue in a short-term basis (10s after the shock) and a long-term basis (2-5 min post-cardioversion) to study the transient and sustained effects, respectively. ST-segment changes (post-shock - pre-shock, post-cardioversion - pre-cardioversion) will be compared between the two defibrillators.
Defibrillator Safety - the rate of patients with elevated biochemical markers | 12 hours after CVS +/- 4 hours
  The rate of patients with elevated biochemical markers for myocardial necrosis including CK-MB and hsTnI 12 hours after the cardioversion procedure. All blood test are done by hospital clinic of clinical laboratory. Elevation above upper limit of normal for CK-MB and above 99 percentile for hsTnI will be compared between the two defibrillators.

CONTACTS AND LOCATIONS:
Overall Officials: Elina G Trendafilova, MD, Principal Investigator — Head of ICCU, NHH
Locations (1):
- University National Heart Hospital, Sofia, Bulgaria

REFERENCES:
- [Derived] Trendafilova E, Dimitrova E, Didon JP, Krasteva V. A Randomized Comparison of Delivered Energy in Cardioversion of Atrial Fibrillation: Biphasic Truncated Exponential Versus Pulsed Biphasic Waveforms. Diagnostics (Basel). 2021 Jun 17;11(6):1107. doi: 10.3390/diagnostics11061107. PMID 34204498